CLINICAL TRIAL: NCT06762925
Title: Study on the Efficacy and Mechanism of METTL3 Peptide Inhibitors in Enhancing Anti-tumor Immune Response by Reshaping the Tumor Microenvironment
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20242214
Record Dates: First submitted 2024-11-21; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer; Prostate Cancer; Kidney Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Bladder Cancer
  Interventions: Other: No Interventions
- Prostate Cancer
  Interventions: Other: No Interventions
- Kidney Cancer
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
This study aims to validate the accuracy and clinical value of METTL3 as a biomarker for predicting immune therapy response in patients with urinary tract tumors through observational studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with urinary system tumors through pathological examination;
2. Meet specific clinical stages and surgical treatment standards;
3. Intraoperative tissue resection meets the sample testing standards;
4. The patient is willing to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. Not meeting the specific clinical stage and not receiving surgical treatment;
2. Abnormal mental behavior;
3. Intellectual disability;
4. Age under 18 years old or over 75 years old;
5. Low understanding and communication skills.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with urological tumors
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The expression levels of METTL3 and ANGPTL2 | About a year and a half